CLINICAL TRIAL: NCT02606188
Title: Modified High-flow Nasal Cannula Oxygen in Patients Undergoing Bronchoscopy.
Brief Title: Modified HFNC Oxygen in Patients Undergoing Bronchoscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haichao Li (Other)
Responsible Party: Sponsor-Investigator, Haichao Li, Sponsor-Investigator, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-ke-091
Record Dates: First submitted 2015-11-14; First posted 2015-11-17 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Bronchoscopy,Oxygen
Keywords: Modified High-flow nasal cannula; Bronchoscopy; Oxygen therapy
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified High-flow nasal cannula therapy (Active Comparator): Patients undergoing bronchoscopy are given Modified High-flow nasal cannula oxygen therapy all the time.
  Interventions: Device: Modified High-flow nasal cannula
- Nasal cnnnula therapy (Active Comparator): Patients undergoing bronchoscopy are given nasal cannula oxygen therapy all the time.
  Interventions: Device: nasal cannula

INTERVENTIONS:
Device: Modified High-flow nasal cannula — Modified High-flow nasal cannula
  Arms: Modified High-flow nasal cannula therapy
Device: nasal cannula — Conventional oxygen therap
  Arms: Nasal cnnnula therapy

SUMMARY:
The purpose of this study is to determine whether the Modified High-flow nasal cannula is effective in the oxygen of the patients undergoing bronchoscopy.

ELIGIBILITY:
Inclusion criteria

1. age more than 18 years old;
2. need for bronchoscopy for diagnosis purpose.

Exclusion criteria

1. peripheral arterial pulse oximetry was < 90%
2. platelet count < 60 × 109/L;
3. nasopharyngeal obstruction or blockage.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2015-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients SpO2 < 90% during bronchoscopy | 1 hour

SECONDARY OUTCOMES:
the operation time | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Department of respiratory and critical care medicine,Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Lucangelo U, Vassallo FG, Marras E, Ferluga M, Beziza E, Comuzzi L, Berlot G, Zin WA. High-flow nasal interface improves oxygenation in patients undergoing bronchoscopy. Crit Care Res Pract. 2012;2012:506382. doi: 10.1155/2012/506382. Epub 2012 May 20. PMID 22666567
- [Result] Diab S, Fraser JF. Maintaining Oxygenation Successfully with High Flow Nasal Cannula during Diagnostic Bronchoscopy on a Postoperative Lung Transplant Patient in the Intensive Care. Case Rep Crit Care. 2014;2014:198262. doi: 10.1155/2014/198262. Epub 2014 Nov 13. PMID 25478241
- [Derived] Wang R, Li HC, Li XY, Tang X, Chu HW, Yuan X, Tong ZH, Sun B. Modified high-flow nasal cannula oxygen therapy versus conventional oxygen therapy in patients undergoing bronchoscopy: a randomized clinical trial. BMC Pulm Med. 2021 Nov 14;21(1):367. doi: 10.1186/s12890-021-01744-8. PMID 34775948